CLINICAL TRIAL: NCT02065245
Title: A Phase I/II, Randomized, Blinded and Placebo-controlled Trial to Evaluate the Safety and Potential Efficacy of Allogeneic Human Mesenchymal Stem Cell Infusion in Patients With Aging Frailty
Brief Title: AllogeneiC Human Mesenchymal Stem Cells (hMSC) in Patients With Aging FRAilTy Via IntravenoUS Delivery
Acronym: CRATUS
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Longeveron Inc. (Industry)
Collaborators: The Emmes Company, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 20130646
Record Dates: First submitted 2014-02-14; First posted 2014-02-17 (Estimated); Results first posted 2021-04-27 (Actual); Last update posted 2021-07-14 (Actual); Status verified 2021-07

CONDITIONS: Frailty
Keywords: Aging Frailty; Frailty; Cardiovascular; Stem Cells
MeSH Terms: conditions — Frailty | interventions — Penicillins

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (7):
- Pilot phase - Group 1 (Experimental): Group 1 participants will receive Allogeneic Human Mesenchymal Stem Cells (allo-hMSCs): 20 million allo-hMSCs/kg delivered via peripheral intravenous infusion. Participants in this group have the option to receive an additional 3 infusions of 100million allo-hMSCs/kg per infusion with a 12 to 18 month interval.
  Interventions: Biological: Allogeneic Human Mesenchymal Stem Cells (allo-hMSCs)
- Pilot Phase - Group 2 (Experimental): Group 2 - Allogeneic Human Mesenchymal Stem Cells (allo-hMSCs): 100 million allo-hMSCs/kg delivered via peripheral intravenous infusion. Participants in this group have the option to receive an additional 3 infusions of 100million allo-hMSCs/kg per infusion with a 12 to 18 month interval.
  Interventions: Biological: Allogeneic Human Mesenchymal Stem Cells (allo-hMSCs)
- Pilot Phase - Group 3 (Experimental): Group 3 - Allogeneic Human Mesenchymal Stem Cells (allo-hMSCs): 200 million allo-hMSCs/kg delivered via peripheral intravenous infusion. Participants in this group have the option to receive an additional 3 infusions of 100million allo-hMSCs/kg per infusion with a 12 to 18 month interval.
  Interventions: Biological: Allogeneic Human Mesenchymal Stem Cells (allo-hMSCs)
- Randomized Phase - Group A (Experimental): Group A - Allogeneic Human Mesenchymal Stem Cells (allo-hMSCs): 100 million allo-hMSCs/kg delivered via peripheral intravenous infusion.
  Interventions: Biological: Allogeneic Human Mesenchymal Stem Cells (allo-hMSCs)
- Randomized phase - Group B (Experimental): Group B - Allogeneic Human Mesenchymal Stem Cells (allo-hMSCs): 200 million allo-hMSCs/kg delivered via peripheral intravenous infusion.
  Interventions: Biological: Allogeneic Human Mesenchymal Stem Cells (allo-hMSCs)
- Randomized Phase - Group C (Experimental): Group C - Placebo delivered via peripheral intravenous infusion. Participants in this group have the option to receive one additional infusion of 100million allo-hMSCs/kg with a 12 to 18 month interval.
  Interventions: Biological: Allogeneic Human Mesenchymal Stem Cells (allo-hMSCs); Biological: Placebo
- Addendum B - Antibiotic free cell Group (Experimental): Allogeneic Human Mesenchymal Stem Cells (allo-hMSCs): 100 million penicillin/streptomycin-free allo-hMSCs/kg delivered via peripheral intravenous infusion. Participants in this group have the option to receive an additional 3 infusions of 100million allo-hMSCs/kg per infusion with a 12 to 18 month interval.
  Interventions: Biological: Allogeneic Human Mesenchymal Stem Cells (allo-hMSCs); Biological: Penicillin/Streptomycin-Free Allogeneic Human Mesenchymal Stem Cells (allo-hMSCs)

INTERVENTIONS:
Biological: Allogeneic Human Mesenchymal Stem Cells (allo-hMSCs) — Allogeneic Human Mesenchymal Stem Cells (allo-hMSCs) administered by peripheral intravenous infusion
Biological: Placebo — Placebo administered by peripheral intravenous infusion.
  Arms: Randomized Phase - Group C
Biological: Penicillin/Streptomycin-Free Allogeneic Human Mesenchymal Stem Cells (allo-hMSCs) — Penicillin/Streptomycin-Free Allogeneic Human Mesenchymal Stem Cells (allo-hMSCs) administered by peripheral intravenous infusion.
  Arms: Addendum B - Antibiotic free cell Group

SUMMARY:
The purpose of this study is to look at the safety of treatment with stem cells in patients with Frailty.

ELIGIBILITY:
Inclusion Criteria:

* Provide written informed consent.
* Subjects age greater than or equal to 60 and less than or equal to 95 years at the time of signing the Informed Consent Form.
* Show signs of frailty apart from a concomitant condition as assessed by the Investigator with a frailty score of 4 to 7 using the Clinical Frailty Scale
* Female subjects with an Follicle-stimulating hormone (FSH) equal to or > 25.8 milli-international units (mIU) /mL (milliliter), if not currently on hormone replacement therapy.

Exclusion Criteria:

* Score of less than or equal to 24 on the Mini Mental State Examination (MMSE)
* Inability to perform any of the assessments required for endpoint analysis (report safety or tolerability concerns, perform pulmonary function tests, undergo blood draws, read and respond to questionnaires.
* Active listing (or expected future listing) for transplant of any organ.
* Clinically important abnormal screening laboratory values, including but not limited to: hemoglobin <8 g/dl, white blood cell count <3000/mm3, platelets<80,000/mm3, international normalized ratio (INR) > 1.5 not due to a reversible cause (i.e. Coumadin), aspartate transaminase, alanine transaminase, or alkaline phosphatase > 3 times upper limit of normal, total bilirubin > 1.5 mg/dl.
* Serious comorbid illness that, in the opinion of the investigator, may compromise the safety or compliance of the patient or preclude successful completion of the study. Including, but not limited to: HIV, advanced liver or renal failure, class III/IV congestive heart failure, myocardial infarction, unstable angina, or cardiac revascularization within the last six months, or severe obstructive ventilatory defect.
* Any other condition that, in the opinion of the investigator, may compromise the safety or compliance of the patient or preclude successful completion of the study.
* Be an organ transplant recipient.
* Have a clinical history of malignancy within 5 years (i.e., patients with prior malignancy must be disease free for 5 years), except curatively-treated basal cell carcinoma, squamous cell carcinoma, melanoma in situ or cervical carcinoma if recurrence occurs.
* Have a non-pulmonary condition that limits lifespan to < 1 year.
* Have a history of drug or alcohol abuse within the past 24 months.
* Be serum positive for HIV, hepatitis B Surface Antigen (BsAg) or Viremic hepatitis C.
* Be currently participating (or participated within the previous 30 days) in an investigational therapeutic or device trial.
* Be a female who is pregnant, nursing, or of childbearing potential while not practicing effective contraceptive methods. Female patients must undergo a blood or urine pregnancy test at screening and within 36 hours prior to infusion.
* Have hypersensitivity to dimethyl sulfoxide (DMSO)

Ages: 60 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2014-03-03 (Actual); Primary Completion 2019-10-02 (Actual); Study Completion 2020-10-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joshua M Hare, MD, Principal Investigator — ISCI / University of Miami Miller School of Medicine
Locations (1):
- ISCI/University of Miami Miller School of Medicine, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Golpanian S, DiFede DL, Pujol MV, Lowery MH, Levis-Dusseau S, Goldstein BJ, Schulman IH, Longsomboon B, Wolf A, Khan A, Heldman AW, Goldschmidt-Clermont PJ, Hare JM. Rationale and design of the allogeneiC human mesenchymal stem cells (hMSC) in patients with aging fRAilTy via intravenoUS delivery (CRATUS) study: A phase I/II, randomized, blinded and placebo controlled trial to evaluate the safety and potential efficacy of allogeneic human mesenchymal stem cell infusion in patients with aging frailty. Oncotarget. 2016 Mar 15;7(11):11899-912. doi: 10.18632/oncotarget.7727. PMID 26933813
- [Background] Tompkins BA, DiFede DL, Khan A, Landin AM, Schulman IH, Pujol MV, Heldman AW, Miki R, Goldschmidt-Clermont PJ, Goldstein BJ, Mushtaq M, Levis-Dusseau S, Byrnes JJ, Lowery M, Natsumeda M, Delgado C, Saltzman R, Vidro-Casiano M, Da Fonseca M, Golpanian S, Premer C, Medina A, Valasaki K, Florea V, Anderson E, El-Khorazaty J, Mendizabal A, Green G, Oliva AA, Hare JM. Allogeneic Mesenchymal Stem Cells Ameliorate Aging Frailty: A Phase II Randomized, Double-Blind, Placebo-Controlled Clinical Trial. J Gerontol A Biol Sci Med Sci. 2017 Oct 12;72(11):1513-1522. doi: 10.1093/gerona/glx137. PMID 28977399
- [Background] Golpanian S, DiFede DL, Khan A, Schulman IH, Landin AM, Tompkins BA, Heldman AW, Miki R, Goldstein BJ, Mushtaq M, Levis-Dusseau S, Byrnes JJ, Lowery M, Natsumeda M, Delgado C, Saltzman R, Vidro-Casiano M, Pujol MV, Da Fonseca M, Oliva AA Jr, Green G, Premer C, Medina A, Valasaki K, Florea V, Anderson E, El-Khorazaty J, Mendizabal A, Goldschmidt-Clermont PJ, Hare JM. Allogeneic Human Mesenchymal Stem Cell Infusions for Aging Frailty. J Gerontol A Biol Sci Med Sci. 2017 Oct 12;72(11):1505-1512. doi: 10.1093/gerona/glx056. PMID 28444181
- See also: Interdisciplinary Stem Cell Institute at the University of Miami Miller School of Medicine — http://isci.med.miami.edu

RESULTS

PARTICIPANT FLOW:
Period: Infusion 1
Arm/Group | Pilot Phase - Group 1 | Pilot Phase - Group 2 | Pilot Phase - Group 3 | Randomized Phase - Group A | Randomized Phase - Group B | Randomized Phase - Group C | Addendum B - Antibiotic Free Cell Group
Started | 5 | 5 | 5 | 10 | 10 | 10 | 20
Completed | 5 | 5 | 4 | 10 | 9 | 10 | 19
Not Completed | 0 | 0 | 1 | 0 | 1 | 0 | 1
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Death | 0 | 0 | 1 | 0 | 1 | 0 | 0
Period: Infusion 2
Arm/Group | Pilot Phase - Group 1 | Pilot Phase - Group 2 | Pilot Phase - Group 3 | Randomized Phase - Group A | Randomized Phase - Group B | Randomized Phase - Group C | Addendum B - Antibiotic Free Cell Group
Started | 5 | 5 | 2 | 0 | 0 | 6 | 12
Completed | 5 | 5 | 2 | 0 | 0 | 6 | 11
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Death | 0 | 0 | 0 | 0 | 0 | 0 | 1
Period: Infusion 3
Arm/Group | Pilot Phase - Group 1 | Pilot Phase - Group 2 | Pilot Phase - Group 3 | Randomized Phase - Group A | Randomized Phase - Group B | Randomized Phase - Group C | Addendum B - Antibiotic Free Cell Group
Started | 3 | 5 | 1 | 0 | 0 | 0 | 0
Completed | 2 | 4 | 1 | 0 | 0 | 0 | 0
Not Completed | 1 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 1 | 1 | 0 | 0 | 0 | 0 | 0
Period: Infusion 4
Arm/Group | Pilot Phase - Group 1 | Pilot Phase - Group 2 | Pilot Phase - Group 3 | Randomized Phase - Group A | Randomized Phase - Group B | Randomized Phase - Group C | Addendum B - Antibiotic Free Cell Group
Started | 1 | 2 | 1 | 0 | 0 | 0 | 0
Completed | 1 | 2 | 1 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pilot Phase - Group 1 | Pilot Phase - Group 2 | Pilot Phase - Group 3 | Randomized Phase - Group A | Randomized Phase - Group B | Randomized Phase - Group C | Addendum B - Antibiotic Free Cell Group | Total
Number analyzed (Participants) | 5 | 5 | 5 | 10 | 10 | 10 | 20 | 65
Age, Continuous [Mean (Standard Deviation); unit: years] | 78.8 (5.167) | 75.8 (4.868) | 79.2 (4.024) | 74.6 (7.23) | 75.9 (8.293) | 74.7 (6.75) | 72.75 (8.896) | 75.015 (7.443)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 0 | 2 | 4 | 4 | 4 | 7 | 24
  Male | 2 | 5 | 3 | 6 | 6 | 6 | 13 | 41
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 1 | 1 | 2 | 1 | 5
  Not Hispanic or Latino | 5 | 5 | 5 | 9 | 9 | 8 | 19 | 60
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  White | 5 | 5 | 5 | 10 | 9 | 10 | 20 | 64
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Any Treatment Emergent - Serious Adverse Events (TE-SAEs)
Description: Incidence of any treatment-emergent serious adverse events (SAE), defined as the composite of: death, non-fatal pulmonary embolism, stroke, hospitalization for worsening dyspnea and clinically significant laboratory test abnormalities.
  * Serum chemistry: chloride, bicarbonate, blood urea nitrogen (BUN), creatinine, glucose, calcium, aspartate aminotransferase (AST), alanine aminotransferase (ALT), total bilirubin (fractionate if total >1.5 times normal), alkaline phosphatase, albumin,
  * Hematology (Complete blood count): hemoglobin, hematocrit, platelets, white blood cells (WBC), WBC differential
Time Frame: One Month post infusion
Population: Participants were allowed to opt-in to receive additional infusion based on cohort
Measure: Number; unit: Incidents
Arm/Group | Pilot Phase - Group 1 | Pilot Phase - Group 2 | Pilot Phase - Group 3 | Randomized Phase - Group A | Randomized Phase - Group B | Randomized Phase - Group C | Addendum B - Antibiotic Free Cell Group
Number analyzed (Participants) | 5 | 5 | 5 | 10 | 10 | 10 | 20
Incidents
  Infusion #1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Infusion #2: number analyzed (Participants) | 5 | 5 | 2 | 0 | 0 | 6 | 12
  Infusion #2 | 0 | 0 | 0 |  |  | 0 | 0
  Infusion #3: number analyzed (Participants) | 3 | 5 | 1 | 0 | 0 | 0 | 0
  Infusion #3 | 0 | 0 | 0 |  |  |  |
  infusion #4: number analyzed (Participants) | 1 | 2 | 1 | 0 | 0 | 0 | 0
  infusion #4 | 0 | 1 | 0 |  |  |  |

2. Secondary Outcome: Change in Frailty as Assessed by CHAMPS Questionnaire
Description: Community Healthy Activities Model Program for Seniors (CHAMPS) questionnaire measures duration of exercise-related activities (hours/week). The Duration variable can range from 0 - 399.75 hours per week. Higher scores indicate more activity.
Time Frame: At baseline and 6 month follow-up visit.
Reporting Status: Not Posted

3. Secondary Outcome: Change in Slowing of Mobility as Measured by 4 Meter Gait Speed Test
Description: 4-meter gait speed test measures the time (in seconds) taken to walk a distance of 4 meters. The total score has a range of 1 point - 4 points with the higher score indicating faster walk speed.
Time Frame: At baseline and 6 month follow-up visit.
Reporting Status: Not Posted

4. Secondary Outcome: Change in Slowing of Mobility as Measured by SPPB
Description: Standard Physical Performance Battery (SPPB) Assessment has total score ranging from 0-4 with the higher score indicating better balance.
Time Frame: At baseline and 6 month follow-up visit.
Reporting Status: Not Posted

5. Secondary Outcome: Change in Weight
Description: Change in weight as measured in kilograms (kg).
Time Frame: At baseline and 6 month follow-up visit.
Reporting Status: Not Posted

6. Secondary Outcome: Change in Diminished Hand Grip Strength
Description: Hand grip strength as assessed by a dynamometer. Grip strength is recorded (in mmHg) three times for each hand. The average reading is reported for each hand.
Time Frame: At baseline and 6 month follow-up visit.
Reporting Status: Not Posted

7. Secondary Outcome: Change in Exhaustion as Measured by the MFI Questionnaire
Description: Multi-dimensional Fatigue Inventory (MFI) Questionnaire contains 20 questions with a 5-point scale. The MFI has total score ranging from 20-100 with the higher score indicating less fatigue.
Time Frame: At baseline and 6 month follow-up visit.
Reporting Status: Not Posted

8. Secondary Outcome: Change in Quality of Life (QoL) as Measured by the ICECAP Questionnaire
Description: Investigating Choice Experiences for the Preferences of Older People (ICEpop) Capability measure for Older people (ICECAP) questionnaire has total score ranging from 5-20 with the higher score indicating greater quality of life.
Time Frame: At baseline and 6 month follow-up visit.
Reporting Status: Not Posted

9. Secondary Outcome: Change in Quality of Life (QoL) as Measured by the SF-36 Questionnaire
Description: Short Form (SF)-36 Questionnaire has consists of eight scaled scores, which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale. Lower scores indicate the more disability, and higher scores indicate less disability.
Time Frame: At baseline and 6 month follow-up visit.
Reporting Status: Not Posted

10. Secondary Outcome: Change in Quality of Life (QoL) as Measured by the EQ-5D-3L Questionnaire
Description: EuroQoL (EQ)- 5 Dimension (5D)- 3 levels (3L) Questionnaire has total score ranging from 0-10 for the 5 dimensions. Higher scores indicate better Quality of Life.
Time Frame: At baseline and 6 month follow-up visit.
Reporting Status: Not Posted

11. Secondary Outcome: Change in Quality of Life (QoL) as Measured by the EQ-5D-3L Overall Health Status Scale.
Description: EuroQoL - 5 Dimension - 3 levels (EQ-5D-3L) Overall health status question has a range of 0-100. Higher scores indicate better Quality of Life.
Time Frame: At baseline and 6 month follow-up visit.
Reporting Status: Not Posted

12. Secondary Outcome: Change in Sense of Smell as Measured by UPSIT
Description: University of Pennsylvania Smell Identification Test (UPSIT) smell test booklet has a total score ranging from 0-40 with higher scores indicating better olfaction.
Time Frame: At baseline and 6 month follow-up visit.
Reporting Status: Not Posted

13. Secondary Outcome: Death
Description: Any reported death from any cause.
Time Frame: Up to 12 months.
Reporting Status: Not Posted

14. Secondary Outcome: Change in Ejection Fraction (EF)
Description: Change in dobutamine stress echocardiogram induced ejection fraction
Time Frame: At baseline and 6 month follow-up visit.
Reporting Status: Not Posted

15. Secondary Outcome: Change in Inflammatory Markers Levels
Description: Change in inflammatory markers including C-Reactive Protein (CRP) and Fibrinogen serum samples as measured in mg/L.
Time Frame: At baseline and 6 month follow-up visit.
Reporting Status: Not Posted

16. Secondary Outcome: Change in Inflammatory Markers
Description: Change in inflammatory markers including Interleukin (IL)-6 and Tumor Necrosis Factor (TNF) Alpha from serum samples as measured in pg/mL.
Time Frame: At baseline and 6 month follow-up visit.
Reporting Status: Not Posted

17. Secondary Outcome: Change in Inflammatory Marker D-dimer Levels
Description: Change in inflammatory marker D-Dimer from serum samples as measured in mg/dL.
Time Frame: At baseline and 6 month follow-up visit.
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Up to 6 years
Arm/Group | Pilot Phase - Group 1 | Pilot Phase - Group 2 | Pilot Phase - Group 3 | Randomized Phase - Group A | Randomized Phase - Group B | Randomized Phase - Group C | Addendum B - Antibiotic Free Cell Group
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/5 | 1/5 | 0/10 | 1/10 | 0/10 | 1/20
Serious Adverse Events (participants affected / at risk) | 0/5 | 1/5 | 1/5 | 0/10 | 2/10 | 0/10 | 1/20
Other Adverse Events (participants affected / at risk) | 0/5 | 0/5 | 0/5 | 0/10 | 0/10 | 0/10 | 0/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pilot Phase - Group 1 (N=5) | Pilot Phase - Group 2 (N=5) | Pilot Phase - Group 3 (N=5) | Randomized Phase - Group A (N=10) | Randomized Phase - Group B (N=10) | Randomized Phase - Group C (N=10) | Addendum B - Antibiotic Free Cell Group (N=20)
Stroke (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Upper Respiratory Infection (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Congestive Heart Failure (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Microscopic Hematuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-03-19): https://cdn.clinicaltrials.gov/large-docs/45/NCT02065245/Prot_SAP_000.pdf